CLINICAL TRIAL: NCT04536701
Title: Collaborative Research: Learning and Improving Alzheimer's Patient-Caregiver Relationships Via Smart Healthcare Technology
Brief Title: Learning and Improving Alzheimer's Patient-Caregiver Relationships Via Smart Healthcare Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Virginia (Other); The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Karen Rose, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019B0406
Record Dates: First submitted 2020-08-19; First posted 2020-09-03 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Caregiver Stress Syndrome
Keywords: Alzheimer Disease; Dementia; Caregiving; Smart Health Technology
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Longitudinal descriptive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia/Caregiver Dyad (Experimental): All dementia/caregiver dyads will have in-home acoustic monitoring to classify mood and will be provided mindfulness-based stress reduction recommendations via a smart phone.
  Interventions: Behavioral: Mood Monitoring and Behavioral Recommendation System

INTERVENTIONS:
Behavioral: Mood Monitoring and Behavioral Recommendation System — The purpose of this project is to develop a monitoring, modeling, and interactive recommendation solution (for caregivers) for in-home dementia patient care that focuses on caregiver-patient relationships. This includes monitoring for mood and stress and analyzing the significance of monitoring those attributes to dementia patient care and subsequent behavior dynamics between the patient and caregiver. In addition, novel and adaptive behavioral suggestions will be provided to family caregivers via text messages on project Smart phones at the right moments aimed to help improve familial interactions related to caregiving, which over time should ameliorate the stressful effects of the patient's illness and reduce strain on caregivers.

SUMMARY:
The purpose of this project is to develop a monitoring, modeling, and interactive recommendation solution (for caregivers) for in-home dementia patient care that focuses on caregiver-patient relationships. This includes monitoring for mood and stress and analyzing the significance of monitoring those attributes to dementia patient care and subsequent behavior dynamics between the patient and caregiver. In addition, novel and adaptive behavioral suggestions at the right moments aims at helping improve familial interactions related to caregiving, which over time should ameliorate the stressful effects of the patient's illness and reduce strain on caregivers. The technical solution consists of a core set of statistical learning based techniques for automated generation of specialized modules required by in-home dementia patient care. There are three main technical components in the solution. The first obtains textual content and prosody from voice and uses advanced machine learning techniques to create classification models. This approach not only monitors patients' behavior, but also caregivers', and infers the underlying dynamics of their interactions, such as changes in mood and stress. The second is the automated creation of classifiers and inference modules tailored to the particular patients and dementia conditions (such as different stages of dementia). The third is an adaptive recommendation system that closes the loop of an in-home behavior monitoring system.

DETAILED DESCRIPTION:
The purpose of this project is to develop a monitoring, modeling, and interactive recommendation solution (for caregivers) for in-home dementia patient care that focuses on caregiver-patient relationships. This includes monitoring for mood and stress and analyzing the significance of monitoring those attributes to dementia patient care and subsequent behavior dynamics between the patient and caregiver. In addition, novel and adaptive behavioral suggestions will be provided to family caregivers via text messages on project Smart phones at the right moments aimed to help improve familial interactions related to caregiving, which over time should ameliorate the stressful effects of the patient's illness and reduce strain on caregivers. The technical solution consists of a core set of statistical learning based techniques for automated generation of specialized modules required by in-home dementia patient care. There are three main technical components in the solution. - The first obtains textual content and prosody from voice and uses advanced machine learning techniques to create classification models. This approach not only monitors patients' behavior, but also caregivers', and infers the underlying dynamics of their interactions, such as changes in mood and stress. - The second is the automated creation of classifiers and inference modules tailored to the particular patients and dementia conditions (such as different stages of dementia). - The third is an adaptive recommendation system that closes the loop of an in-home behavior monitoring system.

ELIGIBILITY:
Inclusion Criteria for persons with dementia:

* Females and males
* Age 60-90 years
* Physician documentation of dementia: Alzheimer's disease, vascular, mixed or unspecified type
* Community-dwelling (living in the home)
* Fluent in English

Inclusion criteria for family caregivers:

* Age 21 years or older
* Informal, unpaid caregiver who resides with the care recipient
* Fluent in English
* Functioning home Wifi
* Scoring above a 3 on the Revised Memory and Behavior Problems Checklist, a clinical cut-off point used to determine caregiver stress.

Exclusion Criteria for persons with dementia:

* Presence of acute illness as this could lead to delirium
* Alcohol abuse or dependence within the past 2 years (DSM-IV criteria)
* History of significant psychiatric illness (e.g., schizophrenia).

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Rose, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko E, Rose KM, Gordon KC, Kim S, Gao Y, Wang P, Wijayasingha L, Wang H, Stankovic JA, Wright KD. Feasibility and Acceptability of the Smarthealth Intervention for Dementia Caregivers. A Qualitative Analysis of a Single-Group Pilot Study. J Adv Nurs. 2025 Jun 26. doi: 10.1111/jan.70007. Online ahead of print. PMID 40566925
- [Derived] Rose KM, Coop Gordon K, Schlegel EC, Mccall M, Gao Y, Ma M, Lenger KA, Ko E, Wright KD, Wang H, Stankovic J. Smarthealth technology study protocol to improve relationships between older adults with dementia and family caregivers. J Adv Nurs. 2021 May;77(5):2519-2529. doi: 10.1111/jan.14714. Epub 2021 Feb 11. PMID 33576064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a Memory Care Clinic at a large Midwestern academic institution, through social media and self-referral from January 2021 through December 2023.
Pre-assignment Details: 11 participant dyads (total of 22 participants) completed baseline data collection. 1 dyad withdrew from the study after completing baseline data collection, but did not complete the intervention.
  While all participants were part of a dyad, only caregiver participants completed surveys and are included in the baseline characteristics data and outcome measures. Baseline Characteristics were not collected for patient participants.
Period: Baseline
Arm/Group | Dementia/Caregiver Dyad
Started | 22
Completed | 22
Not Completed | 0
Period: 4 Weeks Post Baseline
Arm/Group | Dementia/Caregiver Dyad
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Caregiver participants only are included in the Baseline Characteristics. Baseline Characteristics were not collected for dementia patient participants.
Arm/Group | Dementia/Caregiver Dyad
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.09 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Education Level - Above High School [Number; unit: participants] | 11
Employed outside of home [Number; unit: participants] | 3
Married [Number; unit: participants] | 7
Veteran Status [Number; unit: participants] | 2
Caregiving hours/day [Mean (Standard Deviation); unit: hours/day] | 21.18 (6.37)
Caregiver duration [Mean (Standard Deviation); unit: months] | 34.82 (20.26)

OUTCOME MEASURES:

1. Primary Outcome: Depression Anxiety Stress Scale (DASS)
Description: The DASS is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress in 3 subscales of 14 items each. The scores of each subscale range from 0-42. These subscales are scored by the addition of the total item scores. Total score is obtained by summing all subscores. Total minimum score: 0; Total maximum score: 126; A higher score indicates higher levels of emotional distress, depression, anxiety and stress.
  Total: Normal - 0-32; Mild - 33-39; Moderate - 40-49; Severe - 50-57; Extremely severe - 58+
  Depression: Normal - 0-9; Mild -10-12; Moderate -13-20; Severe - 21-27; Extremely severe - 28-42
  Anxiety: Normal - 0-6; Mild - 7-9; Moderate -10-14; Severe -15-19; Extremely severe - 20-42
  Stress: Normal - 0-10; Mild - 11-18; Moderate -19-26; Severe - 27-34; Extremely severe - 35-42
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline - Dementia/Caregiver Dyad; 4 Months Post Baseline - Dementia/Caregiver Dyad: All dementia/caregiver dyads will have in-home acoustic monitoring to classify mood and will be provided mindfulness-based stress reduction recommendations via a smart phone.
  Mood Monitoring and Behavioral Recommendation System: The purpose of this project is to develop a monitoring, modeling, and interactive recommendation solution (for caregivers) for in-home dementia patient care that focuses on caregiver-patient relationships. This includes monitoring for mood and stress and analyzing the significance of monitoring those attributes to dementia patient care and subsequent behavior dynamics between the patient and caregiver. In addition, novel and adaptive behavioral suggestions will be provided to family caregivers via text messages on project Smart phones at the right moments aimed to help improve familial interactions related to caregiving, which over time should ameliorate the stressful effects of the patient's illness and reduce strain on caregivers.
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale
  Total | 26.27 (16.46) | 29.10 (30.29)
  DASS-Depressive mood | 8.09 (5.39) | 10 (10.35)
  DASS-Anxiety | 6 (5.25) | 6.5 (9.23)
  DASS-Stress | 12.18 (7.31) | 12.6 (11.74)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Total DASS score reported; Test type: Superiority; p = 0.444, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Depressive Mood DASS score reported; Test type: Superiority; p = 0.8378, t-test, 2 sided
Statistical Analysis 3: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Anxiety DASS score reported; Test type: Superiority; p = 0.4087, t-test, 2 sided
Statistical Analysis 4: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Stress DASS score reported; Test type: Superiority; p = 0.4124, t-test, 2 sided

2. Primary Outcome: Revised Memory and Behavior Problems Checklist (RMBPC)
Description: RMBPC 24-item, caregiver-report of observable behavioral problems in dementia patients AND the caregiver's stress reactions to these disturbances. It provides a total score and 3 subscale scores (memory, depression, and disruptive behaviors) and scores for caregiver reactions.
  Score ranges - Frequency: Total 0-96; Disruptive 0-32; Depressive 0-36; Memory 0-24. Sum items with scores of 0 to 4 on subscales and total. If question score is 9, exclude it from the sum and item count. Sum items for each subscale, compute the mean item score for each subscale by dividing by the number of items included in the sum.
  Score ranges - Reaction Total 1-96; Disruptive 1-36; Depressive 1-36; Memory 1-24. Include only items with frequency scores of 1 to 4 in the reaction scoring. Compute the mean reaction score by summing reaction scores of these items and then dividing by the number of items included in the sum. A higher score indicates worse outcomes.
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale
  Frequency of Symptoms Total | 13.27 (4.22) | 10.9 (5.47)
  Frequency of Disruptive Symptoms | 3.82 (2.60) | 2.4 (2.95)
  Frequency of Depressive Symptoms | 3.09 (2.59) | 2.1 (2.38)
  Frequency of Memory Symptoms | 6.36 (0.92) | 6.4 (0.84)
  Reaction to Symptoms Total | 26.82 (17.35) | 19.6 (21.90)
  Reaction to Disruptive Symptoms | 9.45 (7.50) | 5.5 (7.53)
  Reaction to Depressive Symptoms | 7.27 (8.26) | 5 (8.41)
  Reaction to Memory Symptoms | 10.09 (6.00) | 9.1 (7.19)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Total RMBPC frequency reported; Test type: Superiority; p = 0.0508, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Frequency of disruptive symptoms on RMBP reported; Test type: Superiority; p = 0.026, t-test, 2 sided
Statistical Analysis 3: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Frequency of depressive symptoms on RMBPC reported; Test type: Superiority; p = 0.1861, t-test, 2 sided
Statistical Analysis 4: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Frequency of memory symptoms on RMBPC reported; Test type: Superiority; p = 0.9535, t-test, 2 sided
Statistical Analysis 5: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; RMBPC reaction total is reported; Test type: Superiority; p = 0.0411, t-test, 2 sided
Statistical Analysis 6: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; RMBPC reaction disruptive symptoms is reported; Test type: Superiority; p = 0.0058, t-test, 2 sided
Statistical Analysis 7: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; RMBPC reaction depressive symptoms is reported; Test type: Superiority; p = 0.2527, t-test, 2 sided
Statistical Analysis 8: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; RMBPC reaction memory symptoms; Test type: Superiority; p = 0.3542, t-test, 2 sided

3. Primary Outcome: Change in Caregiver Emotional Reactivity
Description: The 16-item, Difficulties in Emotion Regulation Scale (DERS-16) will be used to measure caregivers' ability to regulate emotions at baseline and end of study. The scale used is the brief version of a theoretically-driven, valid, and reliable self-report tool used to measure difficulties with emotion regulation. The brief version will be more easily administered with the study population and has been shown to be valid and reliable [41]. Minimum score: 16; Maximum score: 80. A higher score indicates higher levels of caregiver emotional reactivity.
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale | 30.55 (11.85) | 34.3 (15.70)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Test type: Superiority; p = 0.3857, t-test, 2 sided

4. Primary Outcome: Five Facet Mindfulness Questionnaire
Description: Five Facet Mindfulness Questionnaire 39-item to measure capacity for five different domains of mindfulness practice at baseline and end of study. The five facets include non-reactivity to the inner experience, non-judgment of the inner experience, acting with awareness, observing, and describing internal states. All items are scored with a scale of 1-5. Some items are marked to be reverse scored. All items are scored and summed then divided by the total in each category by the number of items in that category to get an average category score. Each category is summed to calculate the Total then divided by the number of items to get an average item score for each subscale. A higher score indicates higher levels of caregiver capacity for mindfulness practices and better outcomes.
  Score ranges: Total 1-5; Observing 1-5; Describing 1- 5; Acting with Awareness 1-5; Non-judging 1-5; Nonreactivity 1-5
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale
  Total | 3.48 (0.58) | 3.44 (0.49)
  Observing | 3.43 (0.93) | 3.44 (0.96)
  Describing | 3.83 (0.56) | 3.71 (0.61)
  Acting with Awareness | 3.17 (0.90) | 3.23 (1.14)
  Non-judging | 3.55 (0.91) | 3.58 (0.98)
  Nonreactivity | 3.42 (0.84) | 3.21 (0.77)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; Five Facet Mindfulness Questionnaire (FFMQ) total reported; Test type: Superiority; p = 0.7213, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; FFMQ Observing reported; Test type: Superiority; p = 0.6075, t-test, 2 sided
Statistical Analysis 3: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; FFMQ Describing reported; Test type: Superiority; p = 0.4136, t-test, 2 sided
Statistical Analysis 4: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; FFMQ Acting with Awareness reported; Test type: Superiority; p = 0.8378, t-test, 2 sided
Statistical Analysis 5: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; FFMQ Nonjudging reported; Test type: Superiority; p = 0.7193, t-test, 2 sided
Statistical Analysis 6: Comparison: Baseline - Dementia/Caregiver Dyad vs 4 Months Post Baseline - Dementia/Caregiver Dyad; FFMQ Nonreactivity reported; Test type: Superiority; p = 0.4145, t-test, 2 sided

5. Primary Outcome: Change in Caregiver Strain
Description: Modified Caregiver Strain Index (MCSI): It is a 13-item self-report measure that examines both subjective and objective elements of caregiver strain. The MCSI showed excellent inter-item and test-retest reliability and was correlated in expected directions with relevant criteria [32]. It has excellent reliability and validity, displays adequate clinical sensitivity, has an established cut-off for determining functional/dysfunctional systems, and has been used successfully on a variety of mental health outcomes [28]. We will use a practice tracking worksheet to assess how much the caregivers practice the exercises over the course of the study. Minimum score: 0; Maximum score: 26. High scores indicates higher caregiver strain.
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale | 14.18 (5.58) | 15.1 (6.84)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad; Test type: Superiority; p = 0.5368, t-test, 2 sided

6. Primary Outcome: Family Assessment Device (FAD)
Description: The FAD is a self-report measure that is given as a set of seven subscales measuring a different dimension of family function. Scores for each dimension (problem solving, communication, roles, affective responsiveness, affective involvement, behavior control, and general functioning) are calculated separately as the mean of the items in that subscale. Scored by summing the endorsed responses (1-4) for each subscale (negatively worded statements are reversed) and dividing by the number of items in each scale. A higher score indicates greater levels of family functioning on all subscales
  Score Ranges: Total 1-4; Problem Solving 1-5; Communication 1-4; Roles 1-4; Affective Responsiveness 1-6; Affective Involvement 1-7; Behavior Control 1-4; General Functioning 1-4
Time Frame: Baseline, 4 months
Population: There was 1 participant who did not complete the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Dementia/Caregiver Dyad | 4 Months Post Baseline - Dementia/Caregiver Dyad
Number analyzed (Participants) | 11 | 10
score on a scale
  FAD Total | 2.13 (0.46) | 2.20 (0.59)
  FAD Problem Solving | 2.15 (0.49) | 2.32 (0.73)
  FAD Communication | 2.29 (0.56) | 2.23 (0.49)
  FAD Roles | 2.29 (0.40) | 2.35 (0.72)
  FAD Affective Responsiveness | 2.27 (0.62) | 2.35 (0.76)
  FAD Affective Involvement | 2.08 (0.43) | 2.20 (0.59)
  FAD Behavior Control | 1.82 (0.49) | 1.91 (0.52)
  FAD General Functioning | 2.05 (0.72) | 2.07 (0.77)
Statistical Analysis 1: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Total reported; Test type: Superiority; p = 0.2845, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Problem Solving is reported; Test type: Superiority; p = 0.1386, t-test, 2 sided
Statistical Analysis 3: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Communication is reported; Test type: Superiority; p = 0.7551, t-test, 2 sided
Statistical Analysis 4: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Roles is reported; Test type: Superiority; p = 0.7213, t-test, 2 sided
Statistical Analysis 5: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Affective Responsiveness is reported; Test type: Superiority; p = 0.3233, t-test, 2 sided
Statistical Analysis 6: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Affective Involvement is reported; Test type: Superiority; p = 0.2832, t-test, 2 sided
Statistical Analysis 7: Comparison: Baseline - Dementia/Caregiver Dyad; FAD Behavior Control is reported; Test type: Superiority; p = 0.6831, t-test, 2 sided
Statistical Analysis 8: Comparison: Baseline - Dementia/Caregiver Dyad; FAD General Functioning is reported; Test type: Superiority; p = 0.6075, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events data was collected for the 4 months each participant dyad was actively enrolled in the study.
Description: All adverse events were reported to staff by participants. Adverse events definition concurs with the ClinicalTrials.gov definition.
Arm/Group | Dementia/Caregiver Dyad
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04536701/Prot_000.pdf
  • Informed Consent Form (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT04536701/ICF_001.pdf